CLINICAL TRIAL: NCT06964841
Title: PRIMARY TESTICULAR LYMPHOMA WITH EXTRA-NODAL STOMACH AFFECTATION
Brief Title: PRIMARY TESTICULAR LYMPHOMA
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Huber Díaz Fuentes, PHD, Instituto Mexicano del Seguro Social
Other Study IDs: 982121
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Testicular Lymphoma
Keywords: testis; lymphoma; nodal; stomach
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
742 / 5.000 A 57-year-old male: Denies chronic degenerative, allergic, traumatic, transfusional, or surgical complications. He denies a family history of testicular cancer or abnormalities in testicular descent.

The patient presented with an enlarged right testicle that had been present for 1 month. He saw his family doctor, who prescribed antibiotic and analgesic treatment, without improvement, and was referred to our service. Upon examination, the right testicle was palpable, nontender, slightly enlarged, indurated, with nodulations measuring 0.5 cm in diameter, and free spermatozoa.

The left testicle was normal.

He underwent radical orchiectomy, which revealed renal testicular lymphoma.

DETAILED DESCRIPTION:
A 57-year-old male: Denies chronic degenerative, allergic, traumatic, transfusional, or surgical complications. He denies a family history of testicular cancer or abnormalities in testicular descent.

The patient presented with an enlarged right testicle that had been present for 1 month. He saw his family doctor, who prescribed antibiotic and analgesic treatment, without improvement, and was referred to our service. Upon examination, the right testicle was palpable, non-tender, slightly enlarged, indurated, with nodulations measuring 0.5 cm in diameter, and free spermatozoa.

The left testicle was normal.

He underwent radical orchiectomy, which revealed renal-testicular lymphoma.

On the first postoperative day, the patient began to have stools with malignant cells and discontinuous invasion of the umbilical cord.

He was evaluated by the Gastroenterology department, who indicated the performance of an endoscopy, which revealed a 6 cm bleeding gastric ulcer. A biopsy was taken and a diffuse B-cell lymphoma was detected.

He was evaluated by the Gastroenterology department, who indicated the performance of an endoscopy, which revealed a large lesion.

On the first postoperative day, the patient began to have stools with malignant cells and discontinuous invasion of the umbilical cord.

He was evaluated by the Gastroenterology department, who indicated the performance of an endoscopy, which revealed a large lesion.

The patient continued to have melena and grade IV anemia. He was referred to pathology, where he was found to have OMS. He showed no improvement despite blood transfusions. He died. Immunohistochemistry for both testicular lesions and on the third postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* Patient with testicular lymphoma

Exclusion Criteria:

* Patient without testicular lymphoma

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 57 year old male with testicular lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
Mortality | 3 months
  Describe the mortality in primary testicular lymphoma

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: Yes
anyone who ask via e-mail
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: anytime
Access Criteria: e-mail

REFERENCES:
- [Background] Motyckova M, Vosahlova V, Belada D, Simkovic M, Zak P. [Primary testicular lymphoma]. Vnitr Lek. 2017 Summer;63(6):415-422. Czech. PMID 28840738